CLINICAL TRIAL: NCT03696329
Title: An Open Label, Balanced, Randomized, Two-treatment, Four-period, Two-sequence, Single Dose, Crossover, Fully Replicated Oral Bioequivalence Study of Tetrabenazine Tablets 25 mg of Dr. Reddy's Laboratories Limited, India Comparing With XENAZINE® (Tetrabenazine) Tablets 25 mg of Lundbeck Inc., USA in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Tetrabenazine Tablets 25 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARL/15/420
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetrabenazine Tablets (Experimental): Tetrabenazine Tablets 25 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Tetrabenazine Tablets 25 mg
- Xenazine (Active Comparator): Xenazine Tablets 25 mg of Lundbeck Inc.
  Interventions: Drug: Tetrabenazine Tablets 25 mg

INTERVENTIONS:
Drug: Tetrabenazine Tablets 25 mg
  Other Names: Xenazine

SUMMARY:
This is an open-label, randomized, four-period, two-treatment, two-sequence, balanced, single dose, crossover, oral bioequivalence study in healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, four-period, two-sequence, single dose, crossover, fully replicated oral bioequivalence study of Tetrabenazine Tablets 25 mg of Dr. Reddy's Laboratories Limited, India comparing with XENAZINE® (tetrabenazine) Tablets 25 mg of Lundbeck Inc., USA in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non pregnant female human subjects, age in the range of 18-45 years both inclusive.
2. Body mass index within the range of 18.5 kg/m2- 24.99 kg/m2 extremes included and body weight > 50 kg.
3. Subjects with normal findings as determined by baseline history, physical examination and vital signs examination (blood pressure, pulse rate, respiration rate and axillary temperature).
4. Subjects with clinically acceptable findings as determined by haemogram, biochemistry, urinalysis, 12 lead ECG.
5. Willingness to follow the protocol requirements especially abstaining from xanthine containing food or beverages (chocolates, tea, coffee or cola drinks) or use of grapefruit juice, any alcoholic products, the use of cigarettes and tobacco products for 48.00 hours prior to dosing until after the last blood sample collection in each study period and adherence to food, fluid and posture restrictions.
6. No history of significant alcoholism.
7. No history of drug abuse (benzodiazepines and barbiturates) for the last one month and other illegal drugs for the last 6 months.
8. Non-smokers, ex-smokers and moderate smokers were included. "Moderate smokers are defined as someone smoking 10 cigarettes or less per day, ex-smokers are someone who completely stopped smoking for at least 3 months."
9. Willing to use an acceptable, effective method of contraception.
10. Subject must be literate, able to sign their name, and able to give voluntary written informed consent for the trial
11. Able to read and understand the Informed Consent Form and Medication guide either in its original form (i.e. in English) or translated into a regional language

Exclusion Criteria:

1. Subject is illiterate.
2. Subjects with a history of depression or prior suicide attempts or ideation
3. Known history of hypersensitivity to Tetrabenazine or related drugs.
4. Requiring medication for any ailment having enzyme-modifying activity in the previous 28 days, prior to dosing day.
5. Subjects who have taken prescription medications or over-the-counter products (including vitamins and minerals) within 14 days prior to administration of Investigational Product.
6. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
7. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, haematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
8. Participation in a clinical drug study or bioequivalence study 90 days prior to Period-I dosing of the present study.
9. History of malignancy or other serious diseases.
10. Blood donation 90 days prior to period I dosing of the present study.
11. Subjects with positive HIV tests, HBsAg or Hepatitis-C tests.
12. Found positive in urine test for drug abuse.
13. History of problem in swallowing.
14. Any contraindication to blood sampling.
15. Found positive serum (β) Beta- hCG (Human Chorionic Gonadotropin) test.
16. Lactating women (currently breast feeding).
17. Female subjects not confirming to using birth control measures, from the date of screening until the completion of the study. Abstinence, barrier methods (condom, diaphragm, etc.) are acceptable.
18. Use of hormonal contraceptives either oral or implants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under curve | Pre-dose (within 1 hour prior to dosing), 0.33, 0.67, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 9.00, 12.00, 16.00, 24.00 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vivekananda Murthi, MBBS, Principal Investigator — Accutest Research Laboratories (I) Pvt. Ltd.
Locations (1):
- Accutest Research Laboratories (I) Pvt. Ltd., Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No